CLINICAL TRIAL: NCT06268210
Title: Neoadjuvant Lazertinib With or Without Chemotherapy for Patients With EGFR-mutated Resectable Non-small Cell Lung Cancer (NeoLazer): a Phase II, Randomized, Multi-center Study
Brief Title: Neoadjuvant Lazertinib With or Without Chemotherapy for Patients With EGFR-mutated Resectable Non-small Cell Lung Cancer
Acronym: NeoLazer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Chang Gon Kim, Principal Investigator, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-1546
Record Dates: First submitted 2024-02-08; First posted 2024-02-20 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lazertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients will receive a combination therapy of Lazertinib and Pemed-S + Carboplatin as neoadjuvant treatment before surgery, followed by post-surgery maintenance with Lazertinib at a dosage of 240 mg once daily for a duration of 3 years.
  Dosages:
  Lazertinib: 240 mg once daily (pre-/post-surgery for 3 years) Pemetrexed: 500 mg/m2 every 3 weeks (neoadjuvant therapy for 3 cycles) Carboplatin: AUC5 every 3 weeks (neoadjuvant therapy for 3 cycles)
  Interventions: Drug: Lazertinib+Pemetrexed+Carboplatin
- Comparator (Active Comparator): Lazertinib will be administered at a dosage of 240 mg once daily, both before and after surgery, for a duration of 3 years.
  Interventions: Drug: Lazertinib

INTERVENTIONS:
Drug: Lazertinib+Pemetrexed+Carboplatin — Lazertinib: 240 mg once daily (pre-/post-surgery for 3 years) Pemetrexed: 500 mg/m2 every 3 weeks (neoadjuvant therapy for 3 cycles) Carboplatin: AUC5 every 3 weeks (neoadjuvant therapy for 3 cycles)
  Arms: Experimental
Drug: Lazertinib — Lazertinib will be administered at a dosage of 240 mg once daily, both before and after surgery, for a duration of 3 years.
  Arms: Comparator

SUMMARY:
In the randomized, multicenter Phase II clinical trial, we aim to evaluate the efficacy and safety of Lazertinib monotherapy or the combination of Lazertinib and cytotoxic chemotherapy as neoadjuvant therapy in patients with resectable, treatment-naive EGFR-mutant (exon 19 deletion or exon 21 L858R) non-small cell lung cancer, ranging from clinical stage IB to IIIB. The study is designed to assess the impact on pathological response, as well as effectiveness and safety considerations.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of providing consent, the patient must be an adult aged 19 years or older.
2. Must have histologically or cytologically confirmed completely resectable, non-squamous non-small cell lung cancer (according to AJCC 8th edition, stages IB-IIIB).
3. Complete surgical resection must be deemed feasible based on the investigator's determination and in accordance with local treatment practices. This decision must be verified through the collaboration of a multidisciplinary team, including surgical oncologists, medical oncologists, and radiation oncologists. (Methods of surgical resection: either lobectomy or segmentectomy)
4. Documented presence of EGFR activating mutations (EGFR exon 19 deletion or L858R mutation).
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Adequate and normal organ and bone marrow function, defined as follows:

   Hemoglobin: ≥9.0 g/dL Absolute neutrophil count: ≥1.5 × 10^9/L Platelet count: ≥100 × 10^9/L Serum bilirubin: ≤1.5 x upper limit of normal (ULN) ALT and AST: ≤2.5 x ULN Creatinine clearance: ≥50 ml/min or serum creatinine ≤1.5 × ULN
7. Life expectancy of more than 6 months.
8. Female patients must agree to use appropriate contraceptive methods, should not be breastfeeding, and if of childbearing potential, must have evidence of non-pregnancy through a negative pregnancy test prior to initiation. Effective contraception should be maintained for up to 3 months after the last dose of Lazertinib (6 months for Pemetrexed/Carboplatin).

   Women over 50 years who have discontinued all exogenous hormone therapy and have been amenorrheic for at least 12 months, considered in a "postmenopausal" state.

   Irreversible surgical infertility due to hysterectomy, bilateral oophorectomy, or bilateral tubal ligation; tubal ligation is not allowed.

   Women under 50 years should be considered in a postmenopausal state if they have discontinued all exogenous hormone therapy for at least 12 months, with LH and FSH levels within the postmenopausal range per the testing institution's criteria.
9. Male patients who have not undergone vasectomy must agree to barrier contraception, specifically condom use, and effective contraception and sperm donation are prohibited for up to 3 months after the last dose of Lazertinib (6 months for Pemetrexed/Carboplatin).

Exclusion Criteria:

1. If there is evidence of locally advanced and/or metastatic disease (Stage IIIC-IV).
2. Known positive status for human immunodeficiency virus (HIV).
3. Evidence of severe or uncontrolled active infections, including chronic active hepatitis B and/or C; patients with chronic hepatitis B virus (HBV) with low viral load (HBV DNA ≤ 500 IU/mL or ≤ 2500 copies/mL) can participate if appropriate antiviral therapy can be continued during the treatment period.
4. Evidence of severe or uncontrolled systemic diseases such as uncontrollable hypertension, active bleeding, etc.
5. History of solid organ transplantation.
6. History of interstitial lung disease (ILD) requiring steroid treatment or clinically active ILD.
7. History of malignancies other than non-small cell lung cancer within the past 3 years at the time of the first dose of the investigational drug (exceptions: treated cervical intraepithelial neoplasia, differentiated thyroid cancer without lymph node involvement, non-melanoma skin cancer).
8. Intractable nausea and vomiting, gastrointestinal disorders, or patients for whom oral administration is not feasible, and those deemed to have absorption disorders that may interfere with Lazertinib absorption, with the exception of cases where clinically significant absorption disorders are not present, as determined by the investigator, in patients who have undergone colon resection.
9. Pregnant or lactating women.
10. Any of the following cardiac criteria:

    Average QT interval corrected for heart rate (QTcF) > 470 msec based on three electrocardiogram (ECG) measurements taken with the screening ECG equipment.

    Clinically significant abnormalities in rhythm, conduction, or morphology at rest on ECG, such as complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval > 250 msec.

    Clinically significant heart failure, congenital long QT syndrome, known concomitant drug administration that prolongs the QT interval, or any factors that increase the risk of QTc prolongation or arrhythmias, such as a family history of QTc prolongation or sudden death under the age of 40.
11. Known hypersensitivity to the active or inactive ingredients of Lazertinib or drugs with a similar chemical structure or belonging to the same class.
12. If, in the investigator's judgment, a patient is unlikely to comply with the clinical trial procedures, restrictions, and requirements, and it is determined that the patient should not participate in the clinical trial.
13. Currently participating or planning to participate in any other interventional clinical trial excluding non-interventional clinical trials.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Primary pathological response | After neo adjuvant treatment(3months)
  Primary pathological response refers to the condition where the proportion of viable tumor cells is defined as 10% or less, indicating a substantial reduction in the survival of tumor cells.

SECONDARY OUTCOMES:
Surgical Resection Methods (Segmentectomy or Lobectomy) | After radical surgery(3months)
  Surgical techniques defined by thoracic surgeons based on the extent of surgical resection during radical surgery.
Pathologic Complete Response | After neo adjuvant treatment(3months)
  Absence of detectable residual tumors in pathological findings after neoadjuvant therapy.
Objective Response Rate | After surgery(3months)
  Percentage of patients exhibiting complete response (CR) or partial response (PR) based on RECIST 1.1 criteria from radiological examinations performed prior to surgical treatment.
Event-Free Survival | End of trial(3years)
  Duration encompassing disease progression in situations where surgical treatment has not been carried out following randomization, excluding disease progression leading to surgical exclusion, disease progression or recurrence post-surgical treatment, or death unrelated to the cause.
Disease-Free Survival | End of trial(3years)
  Duration encompassing disease progression, recurrence, or death unrelated to the cause following surgical treatment.
Overall Survival | End of trial(3years)
  Duration from randomization to death unrelated to the cause.
Number of patients with Adverse events according to CTCAE v5.0 | End of trial(3years)
  Evaluation of the safety profile of the protocol treatment summarized in a table for all safety parameters, including:
  * Adverse events according to CTCAE v5.0, including instances leading to treatment interruption, permanent discontinuation, or death.
  * Severe, serious, or specified adverse events.
  * Death.
  * Laboratory parameters, abnormal findings, and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Hye Ryun Kim, Principal Investigator — Severance Hospital
Locations (1):
- Severance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No